CLINICAL TRIAL: NCT00343707
Title: A Double-blind, Triple Dummy, Placebo-controlled, Randomised, Parallel Group Positron Emission Tomography Study to Investigate the Effects of a 8 Week Administration of GW597599 and Paroxetine Either Alone or in Combination on Regional Cerebral Blood Flow During a Public Speaking Test in Subjects Affected by Social Phobia.
Brief Title: PET (Positron Emission Tomography)/Public Speaking Study With A Combination Of 2 Medications In Social Anxiety Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NKP102280
Record Dates: First submitted 2006-06-21; First posted 2006-06-23 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Depressive Disorder and Anxiety Disorders
Keywords: Social Anxiety Disorder; brain imaging; Positron Emission Tomography; antidepressant
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders; Phobia, Social | interventions — vestipitant; Paroxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: vestipitant
Drug: paroxetine
  Other Names: vestipitant

SUMMARY:
This six-arm study is being conducted to measure the effect of a combination of paroxetine and vestipitant on the arousal induced by public speaking in Seasonal Effective Disorder (SAD) patients, using functional brain imaging readouts (i.e., WAT(Wave Analysis Technology) PET(Positron Emission Tomography)), after one or eight weeks of treatment. The effect of paroxetine alone after one or eight weeks of treatment will also be measured.

DETAILED DESCRIPTION:
A double-blind, double dummy, placebo-controlled, randomised, parallel group positron emission tomography study to investigate the effects of a 8 week administration of vestipitant and paroxetine in combination or paroxetine alone on regional cerebral blood flow during a public speaking test in subjects affected by social anxiety disorder.

ELIGIBILITY:
Inclusion criteria:

* Social phobic ambulatory subjects, defined according to DSM-IV criteria.
* Must be capable of giving informed consent and can comply with the study requirements.
* Women of childbearing potential must agree to acceptable method of birth control.

Exclusion criteria:

* Primary diagnosis within the past 6 months of other psychiatric conditions such as major depression or another anxiety disorder.
* Use of medications for a psychiatric condition including herbals in the past 2-12 weeks according to medication type.
* Subjects who, in the investigator's judgement pose a current, serious suicidal or homicidal risk or have made a suicide attempt within the past 6 months.
* Subjects who currently meet or who met within 6 months prior to screening DSM-IV criteria for substance abuse or subjects who currently meet or who met within 6 months prior to screening DSM-IV criteria for substance dependence (other than nicotine).
* Significantly abnormal blood or urine laboratory tests or electrocardiogram (ECG) findings.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2004-11; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
To assess, by mean of Positron Emission Tomography, the degree of regional Cerebral Blood Flow in different brain regions involved in the emotional brain circuit during public speaking task before treatment and after eight weeks of treatment.

SECONDARY OUTCOMES:
To assess symptomatic and physiological measures of anxiety induced by the public speaking task and social anxiety symptoms during eight weeks of treatment. To evaluate safety, tolerability and the effect on sexual function of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Faria V, Ahs F, Appel L, Linnman C, Bani M, Bettica P, Pich EM, Wahlstedt K, Fredrikson M, Furmark T. Amygdala-frontal couplings characterizing SSRI and placebo response in social anxiety disorder. Int J Neuropsychopharmacol. 2014 Aug;17(8):1149-57. doi: 10.1017/S1461145714000352. Epub 2014 Mar 26. PMID 24666527
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: NKP102280 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: NKP102280 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: NKP102280 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: NKP102280 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: NKP102280 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: NKP102280 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register